CLINICAL TRIAL: NCT00236340
Title: DRAINAGE AMNIOTIQUE A LA SERINGUE OU PAR ASPIRATION CONTINUE DANS LES HYDRAMNIOS SYMPTOMATIQUES. ETUDE PROSPECTIVE RANDOMISEE.
Brief Title: Syringe or Continuous Amnioreduction for Symptomatic Polyhydramnios. A Prospective Randomized Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMNIO-2000
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2005-10

CONDITIONS: Polyhydramnios
Keywords: Amniodrainage; Pregnancy; Amniocentesis
MeSH Terms: conditions — Polyhydramnios

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pregnant Women (Other): 47 single foetal pregnancies and 33 twin pregnancies
  Interventions: Device: Syringe aspiration; Device: Wall suction

INTERVENTIONS:
Device: Syringe aspiration — It consists of performing successive aspirations using a 50ml syringe connected to the needle by a flexible tube.
Device: Wall suction — The tubing is connected to the centralized suction system by continuous vacuum, the value of the applied vacuum is 250mmHg

SUMMARY:
To compare the efficiency and maternal and fetal tolerance of two techniques of amnioreduction used in cases of symptomatic second and third trimester polyhydramnios: syringe manual aspiration technique (S group) and continuous suction technique (C group) set to - 250 mmHg

DETAILED DESCRIPTION:
Polyhydramnios is defined as more than 2 liters of amniotic fluid. Ultrasound diagnosis is made either by measurement of a deepest vertical pocket exceeding 8 cm, or by use of an amniotic fluid index (AFI) exceeding 25 cm. Potential complications of polyhydramnios are preterm labor, premature rupture of membranes, altered utero-placental perfusion, and maternal discomfort.

Amniodrainage has become an established technique to improve maternal comfort and reduce the risks of severe polyhydramnios in both singleton and twin pregnancies, decreasing uterine contractility, as well as over-stretching of membranes and uterus. It also acts on the pathological processes of twin to twin transfusion syndrome.

Several techniques are used to reduce symptomatic polyhydramnios. Passive gravitational drainage is long, does not allow to evacuate larger amounts of amniotic fluid and continuous maternal and fetal monitoring is difficult. The standard syringe technique is often a source of discomfort for both the patient and the operator. Continuous aspiration is faster and limits patient's discomfort.

The aim of this study was to compare the efficiency and maternal and fetal tolerance of these two latter techniques of amnioreduction.

A preliminary study permitted to assess the depression value created at the tip of the needle during amniodrainage: the syringe aspiration technique showed large depression variations from 0 to - 300 millimeters of mercury (mmHg). The continuous wall suction was thus chosen to be set to - 250 mmHg: depression at the needle's tip didn't vary during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with abdomen discumfort and ultrasound diagnosis of polyhydramnios (AFI>25cm)
* Single or twin pregnancies

Exclusion Criteria:

* Multiple pregnancy (more than 3 fetuses)
* Maternal history of placental abruptio
* Fetus with IUGR
* Pregnancy complicated with pre-eclampsia
* Unability to give informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
maternal pain (Analogic visual scale) | After drainage

SECONDARY OUTCOMES:
Volume of amniotic fluid drained | After drainage
Duration of the drainage | After drainage
Uterine activity | After drainage
Recording of Foetal Heart Rate | After drainage
Clinical Retroplacental Haematome | After drainage
Histological analysis of the placentas | After drainage

CONTACTS AND LOCATIONS:
Overall Officials: Franck Perrotin, MD PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Andrea Wagner, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Gilles Body, MD PhD, Study Chair — CHU Bretonneau TOURS
Locations (1):
- CHU Bretonneau, Tours, Centre-Val de Loire, France

REFERENCES:
- [Background] Leung WC, Jouannic JM, Hyett J, Rodeck C, Jauniaux E. Procedure-related complications of rapid amniodrainage in the treatment of polyhydramnios. Ultrasound Obstet Gynecol. 2004 Feb;23(2):154-8. doi: 10.1002/uog.972. PMID 14770396
- [Background] Jauniaux E, Holmes A, Hyett J, Yates R, Rodeck C. Rapid and radical amniodrainage in the treatment of severe twin-twin transfusion syndrome. Prenat Diagn. 2001 Jun;21(6):471-6. doi: 10.1002/pd.96. PMID 11438952
- [Background] Elliott JP, Sawyer AT, Radin TG, Strong RE. Large-volume therapeutic amniocentesis in the treatment of hydramnios. Obstet Gynecol. 1994 Dec;84(6):1025-7. PMID 7970458
- [Background] Dolinger MB, Donnenfeld AE. Therapeutic amniocentesis using a vacuum bottle aspiration system. Obstet Gynecol. 1998 Jan;91(1):143-4. doi: 10.1016/s0029-7844(97)00584-x. PMID 9464739